CLINICAL TRIAL: NCT05466383
Title: Screening and Intervention for Adolescent Idiopathic Scoliosis in Haikou, Hainan Province, China
Brief Title: Screening and Intervention for AIS in Haikou, Hainan Province, China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chaoyin Jiang (Other)
Responsible Party: Sponsor-Investigator, Chaoyin Jiang, Professor, Shanghai 6th People's Hospital
Organization: Shanghai 6th People's Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GTYN2022001
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: AIS
MeSH Terms: interventions — Exercise; Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- recommend exercise - perference exercise (Active Comparator)
  Interventions: Behavioral: Exercise
- recommend exercise - perference brace (Active Comparator)
  Interventions: Device: Brace
- recommend exercise - perference observation (No Intervention)
- recommend brace - perference brace (Active Comparator)
  Interventions: Device: Brace
- recommend brace - perference exercise (Active Comparator)
  Interventions: Behavioral: Exercise
- recommend brace - perference observation (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — Exercise rehabilitation with Schroth method
  Arms: recommend brace - perference exercise; recommend exercise - perference exercise
Device: Brace — Wear an orthopedic brace
  Arms: recommend brace - perference brace; recommend exercise - perference brace

SUMMARY:
This is a single-center, prospective, non-randomized, open-label, interventional, real-world study. The mild/moderate AIS patients will be recruited through screening of 250,000 primary and secondary school students in Haikou, Hainan Province. The patients will be treated with different non-surgical interventions (exercise intervention or brace intervention) according to the physician's recommendations and the patient's intention. Patients will be followed up for 36 months to evaluate the effectiveness and safety of non-surgical interventions in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. 9 years ≤ age ≤ 16 years
2. Diagnosis of AIS
3. 10°≤Cobb's angle<45°
4. Signed informed consent form

Exclusion Criteria:

1. With other developmental disorders, musculoskeletal disorders, nerve disorders, infection disorders, mental disorders, and other disorders
2. Obvious deformity of lower limbs and(or) feet
3. Previous or ongoing treatment of AIS
4. Difficulty to read, understanding, and complete the study questionnaires
5. Any criteria, which, in the opinion of the investigator, suggest that the subject would not be compliant with this study protocol

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Out-of-control rate of treatment | 36 months
  Among the patients with skeletal immaturity (Risser's sign 0, 1, 2), out-of-control rate of treatment at the follow-up to 36 months or at skeletal maturity during the trial (i.e., 4° for female Risser's sign or 5° for male Risser's sign). Out-of-control rate of treatment is defined as either: Cobb angle progression >5°, or Cobb angle ≥45°, or the physician recommends or already has enhanced the intervention regimen (i.e., no intervention change to exercise intervention, no intervention change to brace intervention, or exercise intervention change to brace intervention).

SECONDARY OUTCOMES:
Change in SRS-22 score from baseline over time | at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment
  Change in quality of life (SRS-22 score) from baseline at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment compared with those before treatment
Change in vital capacity from baseline over time | at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment
  Change in vital capacity from baseline at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment compared with those before treatment.
Change in plantar pressure from baseline over time | at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment
  Change in plantar pressure from baseline at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months after treatment compared with those before treatment.
Change in gait from baseline over time | at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment
  Change in gait from baseline at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment compared with those before treatment
Correlation between the treatment compliance and the out-of-control rate of treatment | 36 months
  Correlation between the treatment compliance (average daily duration of treatment for scoliosis) and the out-of-control rate of treatment
Correlation between the skeletal maturity at baseline and the out-of-control rate of treatment | 36 months
  Correlation between the skeletal maturity (Risser's sign) at baseline and the out-of-control rate of treatment
Correlation between the Cobb's angle at baseline and the out-of-control rate of treatment | 36 months
  Correlation between the Cobb's angle at baseline and the out-of-control rate of treatment
Correlation between the immediate correction and the out-of-control rate of treatment | 36 months
  Correlation between the immediate correction [(the baseline of Cobb angle - Cobb angle immediately after wearing the brace)/the baseline of Cobb angle] and the out-of-control rate of treatment
The incidence of adverse events | 36 months
  The incidence of adverse events for the intervention
The change in Cobb angle from baseline over time | 36 months
  The change in Cobb angle from baseline at 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months after treatment compared with those before treatment
Correlation between the treatment compliance and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the treatment compliance (average daily duration of treatment for scoliosis) and the change in 36-month Cobb angle from baseline
Correlation between the skeletal maturity at baseline and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the skeletal maturity (Risser's sign) at baseline and the change in 36-month Cobb angle from baseline
Correlation between the immediate correction and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the immediate correction [(the baseline of Cobb angle - Cobb angle immediately after wearing the brace)/the baseline of Cobb angle] and the change in 36-month Cobb angle from baseline
Correlation between the Cobb's angle at baseline and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the Cobb's angle at baseline and the change in 36-month Cobb angle from baseline

OTHER OUTCOMES:
Correlation between the age and the out-of-control rate of treatment | 36 months
  Correlation between the patient's age and the out-of-control rate of treatment
Correlation between the BMI at baseline and the out-of-control rate of treatment | 36 months
  Correlation between the patient's BMI (kg/m^2) at baseline and the out-of-control rate of treatment
Correlation between the type of AIS and the out-of-control rate of treatment | 36 months
  Correlation between the type of AIS and the out-of-control rate of treatment
Correlation between the types of braces and the out-of-control rate of treatment | 36 months
  Correlation between the types of braces and the out-of-control rate of treatment
Correlation between the average time spent doing homework per day at baseline and the out-of-control rate of treatment | 36 months
  Correlation between the average time (hours) spent doing homework per day at baseline and the out-of-control rate of treatment
Correlation between the vitamin D content at baseline and the out-of-control rate of treatment | 36 months
  Correlation between the serum 25(OH)D (nmol/L) at baseline and the out-of-control rate of treatment
Correlation between the average time spent doing outdoor exercise after school per day at baseline and the out-of-control rate of treatment | 36 months
  Correlation between the average time (hours) spent doing outdoor exercise after school per day at baseline and the out-of-control rate of treatment
Correlation between the age and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the patient's age and the change in 36-month Cobb angle from baseline
Correlation between the BMI at baseline and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the patient's BMI (kg/m^2) at baseline and the change in 36-month Cobb angle from baseline
Correlation between the type of AIS and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the type of AIS and the change in 36-month Cobb angle from baseline
Correlation between the types of braces and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the types of braces and the change in 36-month Cobb angle from baseline
Correlation between the average time spent doing homework per day at baseline and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the average time (hours) spent doing homework per day at baseline and the change in 36-month Cobb angle from baseline
Correlation between the vitamin D content at baseline and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the serum 25(OH)D (nmol/L) at baseline and the change in 36-month Cobb angle from baseline
Correlation between the average time spent doing outdoor exercise after school per day at baseline and the change in 36-month Cobb angle from baseline | 36 months
  Correlation between the average time (hours) spent doing outdoor exercise after school per day at baseline and the change in 36-month Cobb angle from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Haikou orthopedic and diabetes hospital, Haikou orthopedic and diabetes hospital of Shanghai Sixth People's Hospital, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: No